CLINICAL TRIAL: NCT04119934
Title: Personalized Biomedical Risk Assessment for Smoking Cessation in Chronic Obstructive Pulmonary Disease
Brief Title: Personalized Smoking Cessation Infographic in COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-231
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Smoking Cessation
Keywords: Chronic obstructive pulmonary disease; COPD; smoking cessation; smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control - None: A retrospective chart review will assess physician/NP behaviour (rates of smoking cessation counselling and prescription of smoking cessation pharmacotherapy) in the one-year pre-intervention period.
- Intervention - Smoking cessation infographic: Throughout the intervention period, the personalized smoking cessation infographic will be provided to physicians/NPs (for eligible patients). Chart review will be conducted for the patient's physician/NP within a three-month window of receiving the infographic to assess outcomes.
  Interventions: Behavioral: Smoking Cessation Intervention Tool

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention Tool — A personalized smoking cessation infographic is provided to the physician/NP alongside the patient's regular spirometry report.
  Groups: Intervention - Smoking cessation infographic

SUMMARY:
This study assesses the effect of a personalized smoking cessation infographic on physician smoking cessation counseling rates and smoking cessation pharmacotherapy prescription rates. The study assesses the difference in physician behaviour using an interrupted time series analysis (one-year pre vs. one-year post-intervention). General practitioners, nurse practitioners and respirologists who refer eligible patients (COPD, active smoking) for spirometry at the St. Michael's Hospital Pulmonary Function Lab will receive the infographic. This is a quality improvement initiative.

The smoking cessation infographic uses individualized patient data (height, weight, sex, baseline FEV1, etc.) to produce a personalized lung function decline prediction over the next 15 years.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) affects 11.8% of adult Ontarians, remains the leading cause of hospitalization in Canada, and cost the Canadian economy $770 million in 2010. Smoking cessation reduces mortality and improves quality of life in COPD, and also reduces the risk of developing stroke, coronary heart disease, and several types of cancer. Despite this evidence, 45% of patients with COPD continue to smoke.

Previous trials have demonstrated that even brief smoking cessation advice offered by a physician can increase quit rates, with intensive interventions proving additionally effective. Despite this, only 37% of US and 54% of Canadian smokers who had a visit with a physician during the prior year had been advised to quit smoking. Barriers and enablers underlying this care gap are multi-fold. At the patient level, barriers to quitting include accessibility of appropriate therapy, low expectations of quit success (self-efficacy) and low expectations of risk mitigation by quitting (outcome expectancy). Enablers include easily available therapy, knowledge of ongoing smoking effects, and motivation to quit for personal gain. For clinicians, barriers to providing smoking cessation advice include perceived lack of cessation counseling skills (self-efficacy), lack of time, memory (forgetting to do it), and concerns about harming the doctor-patient relationship. Enablers include reminders to provide cessation advice and improved outcome expectancy (a belief that their patients have a reasonable chance of quitting).

Among different lung function metrics, forced expiratory volume in one second (FEV1) is the best validated metric for quantifying the degree of lung function impairment and is used to define disease severity. Our group previously developed and validated a prediction tool that uses individual patient characteristics to predict a personalized rate of future FEV1 decline. Considering the barriers and enablers to effective smoking cessation interventions noted above, our team then designed a smoking cessation intervention centered on this lung function decline calculator. Given that smoking is a modifiable variable that affects the rate of lung function decline, we translated the original calculator into a clinical infographic which quantitatively demonstrates the consequences of quitting versus continuing smoking on lung function and its correlated patient-relevant outcomes, for each individual patient (i.e. a personalized biomedical risk assessment). This approach was informed by previous studies demonstrating the promise of biomedical risk assessment (the process of giving smokers feedback on the physical effects of smoking using physiological measurements) and tailored educational materials for smoking cessation. Such tools can enhance smoking cessation consultations, particularly when educational material is in a visual format. We first designed a prototype tool according to best infographic design and content evidence and then conducted a series of iterative 2-hour moderated focus groups with 4-5 COPD patient participants per group and semi-structured 1-on-1 interviews with respirologists, until saturation of themes [4 focus groups (20 participants), 4 interviews]. In a rapid cycle design process, we made changes to tool content and format after each focus group and interview, based on qualitative analysis of feedback.

This infographic is designed for clinicians to use as a facilitator for smoking cessation intervention delivery with their patients. It demonstrates expected FEV1 decline with and without smoking cessation, and corresponding patient-relevant morbidities (page 1), and provides clinicians with guidance for smoking cessation pharmacotherapy prescriptions (page 2). With this project, we seek to evaluate this tool in real-world practice to determine implementation feasibility and preliminary impact. The tool will not only act as a prompt for clinicians to provide smoking cessation counseling, but also serves to improve their self-efficacy and to enhance outcome expectancy with respect to smoking cessation advice. In turn, it provides patients with a personalized analysis of the future impact of their smoking and the benefit of a quit, with a goal of enhancing motivation to quit.

ELIGIBILITY:
Eligible clinicians will include respirologists, general practitioners and nurse practitioners who refer patients for spirometry testing at the St. Michael's Hospital Pulmonary Function Lab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of clinicians in primary care and hospital settings in Toronto, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible, smoking patients with COPD who receive a smoking cessation counselling intervention | 12 months, broken into individual time series periods
  Using prospective chart review, we will assess the proportion of smoking patients with COPD who receive or are referred to a smoking cessation intervention at or after the index visit, in each analysis period
Proportions of eligible, smoking patients with COPD who are prescribed or recommended smoking cessation pharmacotherapy | 12 months, broken into individual time series periods
  Using prospective chart review, we will assess the proportion of smoking patients with COPD who are prescribed or recommended smoking cessation pharmacotherapy at or after the index visit, in each analysis period

SECONDARY OUTCOMES:
Changes in respiratory medication prescriptions for eligible, smoking patients with COPD | 12 months, broken into individual time series periods
  Chart review will qualitatively record changes in respiratory medication prescriptions in all visits at or after the index visit, in each analysis period. We will include "on treatment" analyses for relevant outcomes (assessing outcomes in situations where patients a) successfully received the infographic; and b) situations where providers utilized the infographic). We will also analyze and adjust outcomes by provider characteristics (type, site, etc.) if event numbers are sufficient.
Changes in recommendations for non-pharmacotherapy smoking cessation strategies for eligible, smoking patients with COPD | 12 months, broken into individual time series periods
  Chart review will qualitatively record changes in recommendations for non-pharmacotherapy smoking cessation strategies in all visits at or after the index visit, in each analysis period.
Smoking cessation billing code changes for eligible, smoking patients with COPD. | 12 months, broken into individual time series periods
  Chart review will assess billing codes used for smoking cessation in all visits at or after the index visit, in each analysis period. We will include "on treatment" analyses for relevant outcomes (assessing outcomes in situations where patients a) successfully received the infographic; and b) situations where providers utilized the infographic). We will also analyze and adjust outcomes by provider characteristics (type, site, etc.) if event numbers are sufficient.
Smoking cessation rates for smoking patients with COPD seen a minimum of 6 months after the index visit, in each analysis period. | 6 months
  Chart review will assess for documentation of smoking cessation in all visits at or after the index visit, in each analysis period.
Smoking reduction rates for smoking patients with COPD seen a minimum of 6 months after the index visit, in each analysis period. | 6 months
  Chart review will assess for documentation of smoking reduction in all visits at or after the index visit, in each analysis period. We will include "on treatment" analyses for relevant outcomes (assessing outcomes in situations where patients a) successfully received the infographic; and b) situations where providers utilized the infographic). We will also analyze and adjust outcomes by provider characteristics (type, site, etc.) if event numbers are sufficient.
Changes in number of spirometry referrals for COPD or query COPD (in smokers and non-smokers) | 12 months, broken into individual time series periods
  A review of the pulmonary function lab visits in each analysis period will assess whether there was an increase in the number of spirometry referrals from the enrolled physicians, and all physicians.
Tool uptake | 12 months
  Chart review will look for evidence of tool use with the patient at the visit in all visits at or after the index visit, in the intervention period.
Qualitative and quantitative user feedback for the tool | 12 months
  Exclusively throughout the intervention, electronic questionnaires and telephone interviews will be solicited to assess user feedback on: barriers/enablers to use, feasibility, effect on workflow, perceived usability, quality and impact on smoking cessation counseling delivery and effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anthonisen NR, Skeans MA, Wise RA, Manfreda J, Kanner RE, Connett JE; Lung Health Study Research Group. The effects of a smoking cessation intervention on 14.5-year mortality: a randomized clinical trial. Ann Intern Med. 2005 Feb 15;142(4):233-9. doi: 10.7326/0003-4819-142-4-200502150-00005. PMID 15710956
- [Background] Chapman KR, Bourbeau J, Rance L. The burden of COPD in Canada: results from the Confronting COPD survey. Respir Med. 2003 Mar;97 Suppl C:S23-31. doi: 10.1016/s0954-6111(03)80022-7. PMID 12647940
- [Background] Schuster MA, McGlynn EA, Brook RH. How good is the quality of health care in the United States? 1998. Milbank Q. 2005;83(4):843-95. doi: 10.1111/j.1468-0009.2005.00403.x. No abstract available. PMID 16279970
- [Background] Zafari Z, Sin DD, Postma DS, Lofdahl CG, Vonk J, Bryan S, Lam S, Tammemagi CM, Khakban R, Man SFP, Tashkin D, Wise RA, Connett JE, McManus B, Ng R, Hollander Z, Sadatsafavi M. Individualized prediction of lung-function decline in chronic obstructive pulmonary disease. CMAJ. 2016 Oct 4;188(14):1004-1011. doi: 10.1503/cmaj.151483. Epub 2016 Aug 2. PMID 27486205
- [Background] Voncken-Brewster V, Tange H, de Vries H, Nagykaldi Z, Winkens B, van der Weijden T. A randomized controlled trial evaluating the effectiveness of a web-based, computer-tailored self-management intervention for people with or at risk for COPD. Int J Chron Obstruct Pulmon Dis. 2015 Jun 8;10:1061-73. doi: 10.2147/COPD.S81295. eCollection 2015. PMID 26089656
- See also: Statistics Canada. Canadian Tobacco Use Monitoring Survey (CTUMS): Detailed Information from February to June 2006 — http://www23.statcan.gc.ca/imdb/p2SV.pl?Function=getSurvey&Id=30140